CLINICAL TRIAL: NCT02474056
Title: The Impact of the Fluid Resuscitation on the Venous Volume and Flow Characteristics in Hypovolemic Shock
Status: Withdrawn | Type: Observational
Why Stopped: The researcher couldnt handle it
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Kopelman doron, Cheif of Surgery department B, HaEmek Medical Center, Israel
Other Study IDs: 0018-09-EMC; 0018-09--EMC
Record Dates: First submitted 2015-06-14; First posted 2015-06-17 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: the Study Focuses on the Subgoup of Patients With Decreased Effective Blood Volume eg. Trauma Surgical and Non Surgical Patients
Keywords: decreased blood volume vein volume flow ultrasound exam

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (3):
- trauma patients: patients with decreased blood volume
- surgical patients: patients with decreased blood volume
- non surgical patients: patients with decreased blood voloume

SUMMARY:
We hypothesis that in various situation when the effective blood volume decreased the venous volume flow characteristics change according to the fluid resuscitation

DETAILED DESCRIPTION:
Patients with clinical signs of loss of the effective blood volume will undergo ultrasound examination of several major veins. The purpose of this examination is to determine vein volume(size) and flow. The ultrasound examination will be done before fluid resuscitation, after fluid administration,and three days after admission

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* decreased effective blood volume
* Systolic blood pressure < 100
* Pulse rate > 110

Exclusion Criteria:

* age <18 years old
* pregnancy
* patient requires urgent surgical intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted at haemek medical center
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
blood volume | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Doron Kopelman, Md, Principal Investigator — haemek medical center
Locations (1):
- Haemek Medical Center, Afula, Israel